CLINICAL TRIAL: NCT03707873
Title: Effect of Targeted Education for Atrial Fibrillation Patients
Acronym: AF-EduCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hein Heidbuchel, Professor Doctor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-EduCare / EC 18/12/171; T002917N (Other Grant/Funding Number: Fund for Scientific Research Flanders (FWO) as Applied Biomedical Research with a Primary Social finality (TBM))
Record Dates: First submitted 2018-10-02; First posted 2018-10-16 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Atrial Fibrillation and Flutter
Keywords: Education
MeSH Terms: conditions — Atrial Fibrillation | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: AF patients will be divided in three groups: one group will have in-person education, the second group will have online education and the third group will receive standard AF care. Cardiovascular outcomes will be compared between these groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person education (Experimental): Education will be given on a regular basis via predefined consultation visits. Medication adherence (oral anticoagulation) will also be measured using a special cap that fits on a medication bottle. If adherence is low, the patient will get additional feedback when he does not take this medication as prescribed.
  Interventions: Other: Education
- Online education (Experimental): Education will be given on a regular basis via a special designed online platform. Medication adherence (oral anticoagulation) will also be measured using a special cap that fits on a medication bottle. If adherence is low, the patient will get additional feedback when he does not take this medication as prescribed.
  Interventions: Other: Education
- Standard Care (No Intervention): This group of AF patients will serve as a control group and no extra focused educational reinforcements will be provided beyond standard care (i.e. information of the treating physician and a brochure).

INTERVENTIONS:
Other: Education — Education + Medication adherence monitoring + Feedback when low adherence
  Arms: In-person education; Online education

SUMMARY:
The aim of this study is to evaluate the effect of targeted in-person and online education on cardiovascular outcomes of AF patients (inpatient and outpatient), compared with standard care. Several other parameters (i.e. knowledge level, quality of life, symptom burden, self-care capabilities, adherence to oral anticoagulation, and an evaluation of the educational efforts) will be studied. Cost-effectiveness and cost-utility will also be investigated.

The main research hypothesis is that individualized education based on the knowledge gaps measured with the JAKQ (Jessa Atrial fibrillation Knowledge Questionnaire) in each individual patient (called 'targeted education') is superior when compared to current AF care, both from an efficacy perspective (evaluated by different outcome measures) and from a cost-effectiveness perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients in whom AF or atrial flutter is diagnosed with an electrocardiogram (12-lead, holter,…)
3. Patients who are capable to sign the informed consent.

Exclusion Criteria:

1. Not able to speak and read Dutch
2. Cognitive impaired (e.g. severe dementia)
3. Life expectancy is estimated to be less than 1 year.
4. Ongoing participation in another clinical trial.
5. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  The occurrence of a composite endpoint of cardiovascular death, cardiovascular hospitalizations (first and recurrent) and unplanned cardiovascular or neurological consultations (first and recurrent).

SECONDARY OUTCOMES:
Patients' knowledge level, assessed by the Jessa Atrial fibrillation Knowledge Questionnaire (JAKQ) | at baseline, 1 month, 3-, 6-, 12- and 18 months and if applicable at 24-, 30- and 36 months or at the end of the study in the intervention groups. In the standard care group at 18 months and if applicable at the end of the study.
  This questionnaire includes 16 knowledge questions: 8 about atrial fibrillation, 5 about oral anticoagulation medication and 3 about vitamine K antagonists or non-vitamin K antagonist oral anticoagulants. A total score between 0% and 100% will be generated in which 100% is the best possible score (all questions are answered correctly).
Patients' quality of life, assessed by the EQ-5D-3L questionnaire and the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire. | at baseline, 3-, 12- and 18 months and if applicable at the end of the study in the intervention groups. In the standard care group at baseline and 18 months and if applicable at the end of the study.
  The EQ-5D-3L descriptive system includes a total of 5 questions for 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression). Each question has 3 levels (no problems, some problems, and extreme problems). The EQ Visual Analogue Scale records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score of 100) and 'Worst imaginable health state' (score of 0). The AFEQT is an atrial fibrillation-specific health-related quality of life questionnaire based on 18 questions in the domain of symptoms, daily activities and treatment concerns. A treatment satisfaction score can be calculated based on 2 additional questions. All questions are rated on a 7 point Likert scale. A scoring key is used to determine an overall AFEQT score and a treatment satisfaction score ranging from 0 to 100. A lower score indicates a worse health-related quality of life.
Patients' symptom burden, assessed by the Leuven ARrhythmia Questionnaire (LARQ). | at baseline, 3-,12- and 18 months and if applicable at the end of the study in the intervention groups. In the standard care group at baseline and 18 months and if applicable at the end of the study.
  The LARQ is based on 6 atrial fibrillation-related symptoms: palpitations, shortness of breath, chest pain, syncope, dizziness and fatigue. For each of these symptoms (except syncope), symptom prevalence, occurrence (frequency, duration, severity), distress, circumstances triggering the symptom, and effect on daily activities are requested. Subscale scores on five domains (symptom frequency, duration, effect on daily activities, severity and distress) are calculated by summing the raw scores and transforming them to a 0-100 scale. Higher scores represent a more pronounced symptom burden.
Patients' self-care capabilities, assessed by the Self-Care Questionnaire (SCQ) | at baseline, 3-,12- and 18 months and if applicable at the end of the study in the intervention groups. In the standard care group at baseline and 18 months and if applicable at the end of the study.
  This questionnaire includes a total of 15 questions. The first 6 questions will be scored on a 1 to 5 Likert scale. 1 is the best score and 5 is the worst score. The other 9 questions measure evolutions of self-care capabilities over time.
Patients' adherence to medication (oral anticoagulation), measured by the Medication Events Monitoring System (MEMS). | monitoring between 0-3 months and 12-15 months and feedback during 3-6 months and 15-18 months in those patients with a low adherence in the intervention groups
Patients' satisfaction of the intervention will be assessed by a study specific Patient Reported Outcome Measure (PROM) questionnaire. | at 12 months in the intervention groups and 18 months in the standard care group.
  The number of questions will depend on the specific group allocation, ranging from a minimum of 4 questions to a maximum of 20 questions. These questions assess patients' satisfaction and opinion about the education provided during the study.
Mortality | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  The occurrence of death will be followed.
(Un)planned hospital admissions | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
Hospital duration | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  The total number of hospitalization days during the follow-up period will be calculated.
(Un)planned cardiovascular and neurological visits | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
Cardiovascular emergency department visits | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
General practitioner visits | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).

OTHER OUTCOMES:
Time investments | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  Time investments will be tracked (e.g. timing of the initiation session, the education sessions, feedback during medication telemonitoring).
Cost-utility analysis | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  A cost-utility analysis will be performed.
Cost-effectiveness analysis | Patients will be followed for a minimum of 18 months (=last included patient) to a maximum of 36 months (=first included patient).
  A cost-effectiveness analysis will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, MD, PhD, Principal Investigator — Universteit Antwerpen
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Edegem
  - Jessa Hospital, Hasselt
  - University Hospitals Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Delesie M, Knaepen L, Dendale P, Vijgen J, Ector J, Desteghe L, Heidbuchel H. Baseline demographics of a contemporary Belgian atrial fibrillation cohort included in a large randomised clinical trial on targeted education and integrated care (AF-EduCare/AF-EduApp study). Front Cardiovasc Med. 2023 Jun 2;10:1186453. doi: 10.3389/fcvm.2023.1186453. eCollection 2023. PMID 37332586